CLINICAL TRIAL: NCT04064580
Title: Analysis of the Capnography Curve Can Allow the Discrimination of Obstructive Patients - Modeling the Capnography Curve
Acronym: CAPNOBST
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7245
Record Dates: First submitted 2019-07-11; First posted 2019-08-22 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-07

CONDITIONS: Respiratory Pathology; Obstructive Syndrome
Keywords: capnography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: diagnostic test — performing a capnography examination

SUMMARY:
Obstructive respiratory diseases such as asthma or COPD are a common reason for emergency room visits. Currently, nasal gill capnography and oxygen saturation measurement (SpO2) are the only two non-invasive means of continuously monitoring a respiratory pathology. To date, Respiratory Functional Explorations (CFE) and more particularly spirometry, are considered as the reference examinations for the diagnosis or monitoring of asthma or COPD. However, physical and physical constraints make their use almost impossible in the context of the emergency with patients presenting to emergencies in respiratory distress, often require oxygen therapy or even non-invasive ventilation. Only pulmonary auscultation can make the diagnosis of acute decompensation of obstructive pathology. This technique is qualitative and imprecise, sometimes leading to a diagnostic uncertainty resulting in delay in taking charge and inappropriate therapy.

Studies have shown a change in the capnography curve in obstructive airway disorder and a strong correlation between some capnography parameters and spirometry parameters such as the Tiffeneau ratio (FEV1 / FVC), suggesting capnography as a simple and effective technique for the diagnosis of obstructive syndrome of patients in emergencies.

ELIGIBILITY:
Inclusion Criteria:

* Major patient male or female
* Patient with respiratory disease with and without obstructive syndrome or patient without respiratory pathology
* Patient requiring spirometry breathing functional exploration
* Subject affiliated to a social health insurance scheme
* Subject able to understand the objectives and the risks related to the research and to give its non opposition

Exclusion Criteria:

* Pregnant and lactating woman
* Patient not affiliated to a social protection scheme
* Subject in exclusion period (determined by previous or current study),
* Impossibility of giving the subject information enlightened (subject in emergency situation, difficulties of understanding the subject, ...)
* Subject under the protection of justice Subject under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Major patient requiring spirometry breathing functional exploration
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-11 (Estimated); Primary Completion 2019-11 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Spirometry measurement | 1 day
  Tiffenau Report Compendium (FEV1 / FVC) and FEV1 for spirometry (gold standard defining presence of obstructive disorder).
  Collection of the capnography curves of each patient allowing in a second time to perform an analysis of the curve by different methods.

CONTACTS AND LOCATIONS:
Locations (1):
- Les Hôpitaux Universitaires de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: Undecided